CLINICAL TRIAL: NCT02138942
Title: Automated Administration of Intravenous Fluids Guided by Dynamic Parameters and Cardiac Output During General Anesthesia: a Pilot Feasibility Study
Brief Title: Automated Administration of Fluids Guided by Dynamic Parameters and Cardiac Output During General Anesthesia
Acronym: Closed Loop
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: non-compliance with the protocol. Arrest requested by the Monitoring Safety committee
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOI/2012/RC-01; 2013-A01186-39 (Other: ANSM)
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia
Keywords: automated vascular filling; Learning Intravenous Resuscitator (LIR); General Surgery; Fluid Therapy
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- The study population (Experimental): See inclusion/exclusion criteria.
  Intervention: LIR
  Interventions: Device: Learning Intravenous Resuscitator (LIR) system

INTERVENTIONS:
Device: Learning Intravenous Resuscitator (LIR) system — The usual patient pathways and recommendations concerning vascular filling remain strictly unchanged in this study. The only thing that differs from usual care is the use of the LIR system to automatically optimize fluid resuscitation during general anesthesia, with continuous supervision by the anesthesiologist present during the entire period of use of the device.

SUMMARY:
The main objective of this study is to demonstrate that the LIR (Learning Intravenous Resuscitator) Closed-Loop Fluid Administration System (hereafter the "LIR system"), a new device for the automated administration of intravenous fluids during major abominal surgery and which allows the reinjection of 250 ml of saline filling (crystalloid or colloid), maintains blood volume at values that are acceptable by the "gold standard", i.e. the anesthetist in charge of the patient.

DETAILED DESCRIPTION:
This is a prospective, bi-center, open "Phase II" type study on a medical device (the LIR system). It is the first trial of the device on humans.

The study, which begins at the signing of consent (made the day before or the day of surgery), ends when the patient leaves the hospital. The LIR system is used on a small population of patients under general anesthesia for the automated administration of intravenous fluids during major abdominal surgery by laparotomy or laparoscopy. Several criteria describing the fluids administered, cardiac output, blood pressure and other parameters will be identified during surgery.

This Phase II study is carried out in two, subsequent stages of size "n1" = 19 and "n" = 42.

Strengthening of security :

* The device will be used under the direct supervision of an anesthesiologist ; he / she can regain control instantly when needed .
* An independent oversight committee will be formed and consulted every 10 patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient will receive general anesthesia for a surgical procedure with the following characteristics: ----- planned abdominal surgery by laparotomy or laparoscopy with a probable duration> 2 hours ----- invasive monitoring of blood pressure ----- administration of crystalloid and colloid (HEA PM <150 kDa)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study: ----- Contraindications to the administration of HES MW <150 kDa ----- Patient classified NYHA> 2 ----- Allergy to HEA
* The patient has a pacemaker
* Surgery with cardiopulmonary bypass
* Surgery on the skull
* Dementia
* Patients with brain pathology (tumor, stroke, Parkinson's disease, ...)
* Patients with a psychiatric disorder, severe depression or psychosis, as well as those receiving antipsychotic treatment
* Limitations concerning the use of respiratory pulse pressure variation: cardiac arrhythmia, spontaneous ventilation, using a volume flow <7 ml / kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
The percentage of fluid (crystalloid or colloid) administration changes per patient performed by the LIR system and approved / accepted by the participating anesthetist. | Day 0, just after surgery
  A change may be non-validated in the following two situations:
  1. Stopping criteria when using the LIR system:
     * malfunction of the device
     * malfunction of the electric syringe (Agilia, Fresenius Kabi, Germany)
     * an abnormality of cardiac output measurement or appearance of a limitation to the use of pulse pressure variation (cardiac arrhythmia, spontaneous ventilation, tidal volume <7 ml / kg of theoretical ideal weight).
  2. Non-validation criteria for fluid administration despite a positive indication by the LIR device: If the answer to the two following questions are both yes, preventing the LIR device from acting is not theoretically justified, and the anesthesiologist must justify stopping the device and record the reason for his/her non-validation of the administration of fluid therapy.
     * The last fill increased cardiac output more than 15%? yes/no
     * The prediction parameter for filling response (pulse pressure variation) indicates vascular filling? yes/no

SECONDARY OUTCOMES:
The number of fluid administration modifications (cristalloid or colloid) performed by the device | Day 0, just after surgery
The number of times the anesthetist in charge of the patient had to intervene with the fluid administration (cristalloid or colloid) system/device. | Day 0, just after surgery
The total volume of HEA and crystalloid infused during the preload optimizations and cardiac output | Day 0, just after surgery
The total amount of crystalloid administered for basic inputs during surgery | Day 0, just after surgery
The total amount of intravenous fluids administered during surgery | Day 0, just after surgery
The mean cardiac output during surgery (liters of blood per minute) | Day 0, just after surgery
The maximum cardiac output during surgery (liters of blood per minute) | Day 0, just after surgery
The minimum cardiac output during surgery (liters of blood per minute) | Day 0, just after surgery
Cardiac output at the end of surgery (liters of blood per minute) | Day 0, just after surgery
The percent % variation in cardiac output during surgery | Day 0, just after surgery
Mean blood pressure during surgery | Day 0, just after surgery
Minimum blood pressure during surgery | Day 0, just after surgery
Maximum blood pressure during surgery | Day 0, just after surgery
% variation in blood pressure during surgery | Day 0, just after surgery
Blood pressure at the end of surgery | Day 0, just after surgery
The percentage of time during which the LIR system maintained an optimal/maximal cardiac output. | Day 0 (at the end of surgery)
  Maximizing cardiac output is defined as the cardiac output value for which a vascular filling (250 ml saline filling) causes less than 10% increase in stroke volume.
The minutes required to achieve maximized cardiac output. | Day 0 (at the end of surgery)
The percentage of time spent in hypotension. | Day 0 (at the end of surgery)
The number of hypotension and hypertension episodes requireing treatment. | Day 0 (just after surgery)
Pulse pressure variation throughout surgery | Day 0 (just after surgery)
Stroke volume throughout surgery | Day 0 (just after surgery)
Stroke volume variation | Day 0 (just after surgery)
Blood lactate | Day 0 (at the end of surgery)
% oxygen saturation of central venous blood | Day 0 (at the end of surgery)
Intraoperative urine output | Day 0 (at the end of surgery)
The occurrence of postoperative complications defined by POSSUM criteria | Day 0 to 3; discharge from the post-intervention monitoring room
Medical device malfunctions: presence/absence | Day 0 to 3; discharge from the post-intervention monitoring room
Admission to ICU; yes/no | Day 0 to 3; discharge from the post-intervention monitoring room
Length of stay in ICU | Day 0 to 3; discharge from the post-intervention monitoring room
Length of hospital stay | Hospital discharge; expected maximum of 28 days
The period between the end of surgery and the recovery of audible gastrointestinal transit (auscultation; gas and stool) | Hospital discharge; expected maximum of 28 days
The period between the end of surgery and the recovery of a liquid diet | Hospital discharge; expected maximum of 28 days
The period between the end of surgery and the resumption of solid food | Hospital discharge; expected maximum of 28 days
The period between the end of surgery and the recovery of intestinal transit | Hospital discharge; expected maximum of 28 days
Creatinemia | Baseline (day 0)
Creatinemia | Day 1
Creatinemia | Day 2
Creatinemia | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Lefrant, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes; Claire Roger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Gricourt Y, Prin Derre C, Demattei C, Bertran S, Louart B, Muller L, Simon N, Lefrant JY, Cuvillon P, Jaber S, Roger C. A Pilot Study Assessing a Closed-Loop System for Goal-Directed Fluid Therapy in Abdominal Surgery Patients. J Pers Med. 2022 Aug 30;12(9):1409. doi: 10.3390/jpm12091409. PMID 36143194